CLINICAL TRIAL: NCT02152046
Title: Retinopathy of Prematurity Screening: Comparison of Pain Using Two Eyelid Retractors
Brief Title: ROP Screening: Comparison of Pain Using Two Eyelid Retractors
Status: Terminated | Type: Observational
Why Stopped: Medical Leave of Absence of the Principal Investigator and study team changes
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00106968; 5823 (Other: Advocate IRB); K5900211 (Other: Advocate Health Care)
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Pain During ROP Exam

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Spring loaded retractor: The Alfonso Eyelid Speculum, newborn size
  Interventions: Procedure: ROP exam with spring loaded retractor
- Screw retractor: Cook Eyelid Speculum, infant size
  Interventions: Procedure: ROP exam with screw retractor

INTERVENTIONS:
Procedure: ROP exam with spring loaded retractor
  Groups: Spring loaded retractor
Procedure: ROP exam with screw retractor
  Groups: Screw retractor

SUMMARY:
Retinopathy of prematurity (ROP) is a major cause of blindness in the world. Initial ocular examinations of infants at risk for ROP are generally conducted between 4-6 weeks postnatally. These exams are vital to protect preterm infants from blindness, but these exams have been shown to cause pain in this population.

Currently two speculums are utilized; the spring loaded Alfonso and the screw loaded Cook eyelid speculum. There is no schedule for who receives which speculum during their exam.

The objective of this study is to evaluate the pain response in the neonatal population, 32 weeks or less, and less than or equal to 1500 grams, undergoing a retractor eye exam for retinopathy of prematurity (ROP) screening.

The primary study aim is to compare the N-PASS pain score between neonates who received a ROP eye exam with the spring loaded Alfonso and the screw loaded Cook eye speculums.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) is a major cause of blindness in the world. It is a vasoproliferative retinopathy that affects premature and low birth-weight infants. Initial ocular examinations of infants at risk for ROP are generally conducted between 4-6 weeks postnatally. These exams are vital to protect preterm infants from blindness, but these exams have been shown to cause pain in this population.

Only two studies alluded to the impact of the eyelid speculum on the pain response and score. Specifically, Hered and Gyland, questioned whether the Alfonso, spring loaded, eyelid lid speculum due to its forceful opening of the eyelid causes more pain. However, no studies were found that included the type of eyelid speculum as a variable of study. In addition, no studies have compared the effect of different eyelid speculums on the pain response.

Currently two speculums are utilized; the spring loaded Alfonso and the screw loaded Cook eyelid speculum. There is no schedule for who receives which speculum during their exam. The investigators team recognizes that the insertion of the eyelid speculum causes a pain response in these infants and would like to determine if there is a difference in the level of that response between the two speculums.

The investigators study will test the difference in pain response when using either a spring loaded eyelid speculum or screw loaded speculum during an ROP exam on premature infants.

The objective of this study is to evaluate the pain response in the neonatal population, 32 weeks or less, and less than or equal to 1500 grams, undergoing a retractor eye exam for retinopathy of prematurity (ROP) screening.

The primary study aim is to compare the N-PASS pain score between neonates who received a ROP eye exam with the spring loaded Alfonso and the screw loaded Cook eye speculums.

ELIGIBILITY:
Inclusion Criteria:

* Neonates who are born at less than or equal to 32 weeks gestation or are less than or equal to 1500 grams birth weight

Exclusion Criteria:

* Neonates who are paralyzed or have a negative pain score
* Neonates undergoing an Avastin injection
* Neonates undergoing a Retcam exam
* Neonates transferred to another unit

Ages: 23 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants, who need an ROP exam based on clinical indication.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2014-06-20 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
N-PASS Score immediately after the second eye | 5 minutes
  With each exam, an N-PASS score will be recorded: just prior to the start of the exam; between each eye; at the end of the exam and every minute for five minutes from the completion of the exam.

SECONDARY OUTCOMES:
time it takes for neonates pain score to return to baseline or up to 5 minutes after the end of the exam | 5 minutes
  Time in seconds will be recorded via stopwatch for the entire eye exam, starting with the insertion of the eyelid speculum in the right eye and concluding when the eyelid speculum is removed from the left eyelid.
Maximum pain score recorded | 5 minutes
  With each exam, an N-PASS score will be recorded: just prior to the start of the exam; between each eye; at the end of the exam and every minute for five minutes from the completion of the exam.

OTHER OUTCOMES:
Bradycardia | 5 minutes
  Episodes of bradycardia will be recorded during the eye exam

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Skopec, RN, BSN, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois, United States

REFERENCES:
- [Background] Hummel P, Lawlor-Klean P, Weiss MG. Validity and reliability of the N-PASS assessment tool with acute pain. J Perinatol. 2010 Jul;30(7):474-8. doi: 10.1038/jp.2009.185. Epub 2009 Nov 19. PMID 19924132
- [Background] Hummel P, Puchalski M, Creech SD, Weiss MG. Clinical reliability and validity of the N-PASS: neonatal pain, agitation and sedation scale with prolonged pain. J Perinatol. 2008 Jan;28(1):55-60. doi: 10.1038/sj.jp.7211861. Epub 2007 Oct 25. PMID 18165830